CLINICAL TRIAL: NCT02716272
Title: A Randomized Phase II Study Evaluating Efficacy and Safety of 2nd or 3rd Line Treatment by Nivolumab Monotherapy or Nivolumab Plus Ipilimumab, for Unresectable Malignant Pleural Mesothelioma (MPM) Patients
Brief Title: Nivolumab Monotherapy or Nivolumab Plus Ipilimumab, for Unresectable Malignant Pleural Mesothelioma (MPM) Patients
Acronym: MAPS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1501
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Mesothelioma
Keywords: mesothelioma; immunotherapy; nivolumab; ipilimumab
MeSH Terms: conditions — Mesothelioma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MONOTHERAPY ARM (Experimental): Nivolumab administered IV over 60 minutes at 3mg/kg every 2 weeks
  Interventions: Drug: Nivolumab
- COMBINATION ARM (Experimental): Nivolumab administered IV over 60 minutes at 3mg/kg every 2 weeks, combined with Ipilimumab administered IV over 90 minutes at 1mg/Kg every 6 weeks
  Interventions: Drug: Nivolumab + Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab administered IV over 60 minutes at 3mg/kg every 2 weeks
  Arms: MONOTHERAPY ARM
Drug: Nivolumab + Ipilimumab — Nivolumab administered IV over 60 minutes at 3mg/kg every 2 weeks, combined with Ipilimumab administered IV over 90 minutes at 1mg/Kg every 6 weeks
  Arms: COMBINATION ARM

SUMMARY:
The sponsor raise the hypothesis that inhibition of immune PD-1+/- CTLA-4 check-point(s) would delay tumor progression in patients with unresectable MPM, experiencing disease progression after one or two lines of chemotherapy including at least first-line with pemetrexed and platinum, without altering significantly the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved diagnosis of unresectable malignant pleural Mesothelioma (MPM)
2. Available (archival and/or fresh) pathological samples for centralized PD-L1 expression assessment by immunohistochemistry
3. Age ≥ 18 years old; male and female
4. ECOG Performance status 0-1
5. Weight loss < 10% during last 3 months
6. Life expectancy > 12 weeks
7. Documented progression of the MPM, assessed by computed tomography (CT) -Scan.
8. Measurable disease, defined as at least 1 lesion (measurable) that can be accurately assessed at baseline by CT-Scan and is suitable for repeated assessment using modified Response Evaluation Criteria in Solid Tumors [RECIST] for pleural mesothelioma (Byrne 2004; Therasse 2006).
9. Previous treatment by 1 or 2 systemic chemotherapy lines (1 line of chemotherapy considered if the patient received ≥2 cycles of this chemotherapy), including at least one line with pemetrexed in combination with platinum agent (i.e. "gold standard chemotherapy in MPM; triplet including bevacizumab also accepted)
10. Written informed consent
11. Patients must have adequate organ function : creatinine clearance > 50 mL/min (Cockcroft formula), Neutrophiles count > 1500/mm3; Platelets > 100 000/mm3 ; Hemoglobin > 9 g/dL; hepatic enzymes < 3N with total bilirubin ≤ 1.5 × ULN (upper limit of normal) except subjects with documented Gilbert's syndrome (≤ 5 × ULN) or liver metastasis, who must have a baseline total bilirubin ≤ 3.0 mg/dL
12. Recovered from all toxicities associated with prior treatment, to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.0) Grade of 0 or 1, except for toxicities not considered a safety risk, such as alopecia or vitiligo
13. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 6 months after the final dose of investigational product. Men receiving nivolumab and who are sexually active with women of childbearing potential will be instructed to adhere to contraception for a period of 31 weeks after the last dose of nivolumab.

Exclusion Criteria:

1. Patients with primitive peritoneal, pericardial, testis or tunica vaginalis mesothelioma
2. Patients with a recent history of other malignancies except adequately treated non-melanoma skin cancer, and curatively treated in-situ cancer. Patients with prostate adenocarcinoma diagnosed less than 5 years could be included in case of localized prostate cancer with good outcome according the Amico classification: ≤ T2a and Gleason Score ≤6 and PSA blood level ≤10 ng/ml, and treated with curative intent (surgery or radiotherapy) without chemotherapy. Patients with history of solid tumors, including adenocarcinoma, treated with curative intent and without any evidence of disease >5 years can be included as well.
3. Brain metastasis, except if surgically resected or treated with stereotaxic radiotherapy with no evolution within the 3 months before inclusion, and asymptomatic patient
4. History of primary immunodeficiency, history of organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Intranasal/inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
6. Live attenuated vaccination administered within 30 days prior to randomization.
7. Known history of interstitial lung disease (asbestosis…) or CT-scan signs of interstitial lung disease.
8. Subjects with an active, known or suspected autoimmune disease, including systemic lupus erythematosis or Wegener's granulomatosis. Subjects with type I diabetes mellitis, or hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, are permitted to enroll.
9. Active or history of inflammatory bowel disease (eg, diverticulitis, colitis, Crohn's), irritable bowel disease, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea. Note that diverticulosis is permitted.
10. Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

    * known prior history of active tuberculosis-disease;
    * known acute or chronic B or C hepatitis by serological evaluation. Patients with serological sequelae of hepatitis (antibodies test serologically positive for virus) without hepatitis could be included.
    * known Human immunodeficiency virus infection.
11. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
12. The last dose of prior chemotherapy or radiation therapy (with the exception of palliative radiotherapy) was received less than 3 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-06-22 (Actual)

PRIMARY OUTCOMES:
Disease Control rate assessed by CT scan | 3-months
  Tumor assessment (modified RECIST1.0 for mesothelioma)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3-months
  NCI CTC AE 4.0
Progression-Free Survival | 3-month
Overall Survival | 3-months
Quality of Life | 3-months
  LCSS ( Lawrence County School System) Scale
prognosis impact of blood biomarkers (exploratory studies) | 3-months
  dosage in blood of numerous biomarkers and analysis of their prognosis impact

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Scherpereel, MD, PhD, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique; Gérard Zalcman, MD, PhD, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (22):
- France (22):
  - Angers - CHU, Angers
  - Avignon - Institut Sainte-Catherine, Avignon
  - CHU, Clermont-Ferrand
  - Dijon - CHU, Dijon
  - Grenoble - CHU, Grenoble
  - Centre Hospitalier - Pneumologie, Le Havre
  - Centre Hospitalier - Pneumologie, Le Mans
  - CHRU Lille - Hopital Calmette, Lille
  - AP-HM Hôpital Nord, Marseille
  - Mulhouse - CH, Mulhouse
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - AP-HP Hôpital Bichat, Paris
  - HCL Lyon Sud, Pierre-Bénite
  - Pontoise - CH, Pontoise
  - Rennes - CHU, Rennes
  - Rouen - CHU, Rouen
  - Centre Etienne Dolet, Saint-Nazaire
  - CHU Strasbourg, Strasbourg
  - Toulon - CHI, Toulon
  - Toulouse - CHU Larrey, Toulouse
  - CHU Tours - Pneumologie, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scherpereel A, Mazieres J, Greillier L, Lantuejoul S, Do P, Bylicki O, Monnet I, Corre R, Audigier-Valette C, Locatelli-Sanchez M, Molinier O, Guisier F, Urban T, Ligeza-Poisson C, Planchard D, Amour E, Morin F, Moro-Sibilot D, Zalcman G; French Cooperative Thoracic Intergroup. Nivolumab or nivolumab plus ipilimumab in patients with relapsed malignant pleural mesothelioma (IFCT-1501 MAPS2): a multicentre, open-label, randomised, non-comparative, phase 2 trial. Lancet Oncol. 2019 Feb;20(2):239-253. doi: 10.1016/S1470-2045(18)30765-4. Epub 2019 Jan 16. PMID 30660609
- See also: Official website — http://www.ifct.fr/index.php/fr/la-recherche/item/2033-ifct-1501-maps2